CLINICAL TRIAL: NCT06446518
Title: A Randomized Control Trial for Assessing Virtual Reality for Perioperative Anxiolysis and Postoperative Pain Modulation in Adolescents Undergoing MIRPE Surgery
Brief Title: Assessing Virtual Reality for Perioperative Anxiolysis in Adolescents Undergoing MIRPE Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University (Other)
Collaborators: Új Nemzeti Kiválóság Program (Unknown)
Responsible Party: Principal Investigator, Agnes Jermendy MD PhD MPH, Professor of Pediatrics, Semmelweis University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NRG 2022/2
Record Dates: First submitted 2024-05-31; First posted 2024-06-06 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-07

CONDITIONS: Pectus Excavatum; Pectus Deformity
MeSH Terms: conditions — Funnel Chest

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VR intervention group (Experimental): On admission, patients are asked to fill out a STAI-T and-S anxiety inventory. Attending investigator will take vital parameters upon admission.
  Patients are asked to use the VR headset a minimum of 1 hour before surgery. Participants are asked to fill out a STAI-S test in the operating room, where physiologic data is collected and timing and dose of medication administered. After surgery, during emergence physiologic data is collected, and attending anesthesiologist fills out the PAED score. Patients are encouraged to use the VR headset after surgery, any time when they feel comfortable.
  Pain using an NRS scale, and vital parameters are monitored postoperative 1, 2, 3, 6, 12 hours (if patient is not sleeping) and in the morning following surgery at 6 and 9 am. A final STAI-S test is filled out by patients in the morning after surgery. Data regarding painkiller demand is collected after surgery.
  Interventions: Device: Virtual reality exposure
- Control group (No Intervention): On admission, patients are asked to fill out a STAI-T and-S anxiety inventory. Attending investigator will take vital parameters upon admission.
  Participants are asked to fill out a STAI-S test in the operating room, where physiologic data is collected and timing and dose of medication administered. After surgery, during emergence physiologic data is collected, and attending anesthesiologist fills out the PAED score.
  Pain using an NRS scale, and vital parameters are monitored postoperative 1, 2, 3, 6, 12 hours (if patient is not sleeping) and in the morning following surgery at 6 and 9 am. A final STAI-S test is filled out by patients in the morning after surgery. Data regarding painkiller demand is collected after surgery.

INTERVENTIONS:
Device: Virtual reality exposure — Assessing immersive virtual reality as a distraction tool in anxiolysis and pain modulation.
  Arms: VR intervention group

SUMMARY:
In this randomized control trial, investigators would like to assess as primary objective the effectiveness of VR in anxiolysis via using State Trait Anxiety- Inventory test various time during the perioperative period with recorded physiologic data. As a secondary objective they are investigating the use of VR in the postoperative period for pain modulation via using pain numeric rating scales (NRS), monitoring physiologic data, and collecting information on painkiller demand of the patients.

DETAILED DESCRIPTION:
This prospective, randomized controlled trial will be conducted with participants from the Paediatric Center, Semmelweis University, a tertiary level health care centre based in Budapest, Hungary. We evaluate the effects of VR immersion on reducing perioperative anxiety and postoperative pain.

Participants will be asked to wear a VR headset for preferably an hour before and after the surgery. Patients will be asked to fill out three anxiety tests meanwhile investigators will record their vital parameters (HR, RR, SpO2, BP): on admission, in the operating room and on the surgical ward on the day after surgery. In the first postoperative day vital parameters, analgesic demand and NRS score will be recorded to follow patients pain status.

Researchers will compare VR group to control group to see if anxiety and pain was different among those who recieved the VR headset.

ELIGIBILITY:
Inclusion Criteria:

* Patient between 13-18 years old
* reported chest deformity (pectus excavatum/ carinatum)
* patients undergoing MIRPE surgery in general anesthesia
* Hungarian fluency
* willing to comply with study procedures.

Exclusion Criteria:

* gross cognitive impairment that would interfere with the ability to consent or complete study procedures.
* Head injury
* Head infection
* Altered mental status (independently from midazolam)
* Scabies or louse
* Dizziness or vertigo
* Blindness or severe vision loss
* Lack of parental/ guardian or patient consent
* Those, who has a head deformity, so VR headset does not fit well

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2022-08-17 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Change in anxiety | 1-2 days
  Anxiety assessed by STAI-S and STAI-T questionnaires level of anxiety will be assessed using the State Trait Anxiety-Inventory. The test is composed of 2 parts: STAI-S (How does the patient feel right now?) and STAI-T (How does the patient feel on average?). Both questionnaires contain 20 questions with answers rating from 1 to 4.

SECONDARY OUTCOMES:
Change in pain and vital parameters | 1-2 days
  Pain assessed by Numerical Pain Rating Scale level of pain will be assessed using the Numerical Pain Rating Scale. The scale is composed of 0 (no pain) to 10 (worst pain imaginable).
  Vital parameters that are monitored during the study are blood pressure, heart rate, peripheral oxygen saturation and respiratory rate.
  Pain will also be followed with analgesic demand per patien during the first postoperative day.

CONTACTS AND LOCATIONS:
Locations (1):
- Paediatric Centre, Semmelweis University, Budapest, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: Yes
All relevant variables, that was collected during the study period will be shared after deidentifying the data.

REFERENCES:
- [Background] Kain ZN, Wang SM, Mayes LC, Caramico LA, Hofstadter MB. Distress during the induction of anesthesia and postoperative behavioral outcomes. Anesth Analg. 1999 May;88(5):1042-7. doi: 10.1097/00000539-199905000-00013. PMID 10320165
- [Background] Kain ZN, Mayes LC, O'Connor TZ, Cicchetti DV. Preoperative anxiety in children. Predictors and outcomes. Arch Pediatr Adolesc Med. 1996 Dec;150(12):1238-45. doi: 10.1001/archpedi.1996.02170370016002. PMID 8953995
- [Background] Klassen JA, Liang Y, Tjosvold L, Klassen TP, Hartling L. Music for pain and anxiety in children undergoing medical procedures: a systematic review of randomized controlled trials. Ambul Pediatr. 2008 Mar-Apr;8(2):117-28. doi: 10.1016/j.ambp.2007.12.005. PMID 18355741
- [Background] Eijlers R, Utens EMWJ, Staals LM, de Nijs PFA, Berghmans JM, Wijnen RMH, Hillegers MHJ, Dierckx B, Legerstee JS. Systematic Review and Meta-analysis of Virtual Reality in Pediatrics: Effects on Pain and Anxiety. Anesth Analg. 2019 Nov;129(5):1344-1353. doi: 10.1213/ANE.0000000000004165. PMID 31136330
- [Background] Esposito C, Autorino G, Iervolino A, Vozzella EA, Cerulo M, Esposito G, Coppola V, Carulli R, Cortese G, Gallo L, Escolino M. Efficacy of a Virtual Reality Program in Pediatric Surgery to Reduce Anxiety and Distress Symptoms in the Preoperative Phase: A Prospective Randomized Clinical Trial. J Laparoendosc Adv Surg Tech A. 2022 Feb;32(2):197-203. doi: 10.1089/lap.2021.0566. Epub 2021 Dec 28. PMID 34962159
- [Background] Buyuk ET, Odabasoglu E, Uzsen H, Koyun M. The effect of virtual reality on Children's anxiety, fear, and pain levels before circumcision. J Pediatr Urol. 2021 Aug;17(4):567.e1-567.e8. doi: 10.1016/j.jpurol.2021.04.008. Epub 2021 Apr 21. PMID 34006462
- [Background] Jung MJ, Libaw JS, Ma K, Whitlock EL, Feiner JR, Sinskey JL. Pediatric Distraction on Induction of Anesthesia With Virtual Reality and Perioperative Anxiolysis: A Randomized Controlled Trial. Anesth Analg. 2021 Mar 1;132(3):798-806. doi: 10.1213/ANE.0000000000005004. PMID 32618627
- [Background] Rumsey N, Harcourt D. Body image and disfigurement: issues and interventions. Body Image. 2004 Jan;1(1):83-97. doi: 10.1016/S1740-1445(03)00005-6. PMID 18089143
- [Background] Casatori L, Pellegrino A, Messineo A, Ghionzoli M, Facchini F, Modesti A, Modesti PA. Differential Influence of Physical Activity on Cardiopulmonary Performance and Stroke Volume Assessed at Cardiopulmonary Exercise Test in Pectus Excavatum: A Pilot Study. Front Physiol. 2022 Feb 3;13:831504. doi: 10.3389/fphys.2022.831504. eCollection 2022. PMID 35185624